CLINICAL TRIAL: NCT05539274
Title: Cervical Carcinoma in Shatby University Hospital and Its Relation to Human Papilloma Virus
Status: Completed | Type: Observational
Sponsor: Hossam Hassan Aly Hassan El Sokkary (Other)
Responsible Party: Sponsor-Investigator, Hossam Hassan Aly Hassan El Sokkary, Associate professor, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: Sokkary11
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Genotype

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cervical cancer group, control group
  Interventions: Diagnostic Test: human papilloma virus testing and genotyping in cervical cancer cases

INTERVENTIONS:
Diagnostic Test: human papilloma virus testing and genotyping in cervical cancer cases — an observational analytical prospective cross-sectional study was managed from July 2019 to July 2022 on 70 cervical cancer patients collected from gyne-oncology unit in Shatby obstetrics and gynecology university hospital of Alexandria medical school after taking a written consent and following approval by Alexandria medical school institutional ethics committee. All patients were subjected to full history taking as age, gravidity, parity, contraceptive history, medical disease, detailed marital history and smoking. Collection of the sample from all cases of the study for human papilloma virus testing and genotyping was done after diagnostic workup and before treatment of the study cases at any time in post-menopausal women and at mid cycles period in premenopausal women by cervical smear using PAP spatula and endocervical brush.

SUMMARY:
incidence of detection of carcinogenic types of human papilloma virus in 60 cases of cervical cancer

ELIGIBILITY:
Inclusion Criteria:

* cervical cancer

Exclusion Criteria:

* none

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: cervical cancer cases
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Detection of human papilloma virus infections and genotyping using real time PCR | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hossam Hassan El Sokkary, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No